CLINICAL TRIAL: NCT07037173
Title: Effect of K-Taping and Yoga Therapy in Postural Correction for Sacroiliac Jointamong Weightlifters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1009
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sacroiliac Joint Dysfunction
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping (Experimental)
  Interventions: Combination Product: Kinesiology Taping
- Yoga Therapy (Experimental)
  Interventions: Combination Product: Yoga Therapy

INTERVENTIONS:
Combination Product: Kinesiology Taping — Elastic therapeutic tape applied over the SiJ region using a standardized protocol. Therapy sessions were supervised and conducted at a rehabilitation center three times per week for six weeks.
  Arms: Kinesiology Taping
Combination Product: Yoga Therapy — A structured yoga program including asanas, pranayama, and mindfulness practices focused on enhancing flexibility, core strength, and posture. conducted at a yoga center
  Arms: Yoga Therapy

SUMMARY:
The study investigates the efficacy of kinesiology taping (K-taping) and yoga therapy- both individually and in combination-in correcting posture and rehabilitating sacroiliac joint (SIJ) dysfunction in weightlifters. SIJ dysfunction, commonly caused by repetitive stress, poor biomechanics, and muscle imbalance, is prevalent among weightlifters and can lead to pain and reduced performance.

DETAILED DESCRIPTION:
While K-taping offers immediate support and proprioceptive benefits, yoga therapy provides long-term improvements through enhanced flexibility, core strength, and body awareness.

This study aims to provide evidence for a more integrated and holistic renabilitation approach for Sacroiliac joint.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40
* Diagnosed with SIJ dysfunction
* Visible postural imbalance
* Willing to participate and provide consent

Exclusion Criteria:

* Spinal/pelvic pathologies (e.g., disc herniation)
* Recent trauma/surgery
* Chronic illnesses (e.g., rheumatoid arthritis)
* Pregnancy
* Allergy to tape or restriction from yoga
* Recent trauma/surgery
* Chronic illnesses (e.g., rheumatoid arthritis)
* Pregnancy
* Allergy to tape or restriction from yoga
* Participation in other clinical trials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 6 Month
  Assesses functional disability; scored 0-100%, higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sehat Medical Complex Hanjarwal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No